CLINICAL TRIAL: NCT06096194
Title: Effect of the Consuption of Vitamin D3-enhanced Eggs on Serum 25-hydroxivitamin D[(25-OH)D3] and Parathyroid Hormone (PTH) in Preschool Children
Brief Title: Vitamin D3-enhanced Eggs in Preschool Children
Acronym: VD3-egg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Mario Flores-Aldana, Mario Flores-Aldana, MD, PhD Nutrition Surveillance, Director, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FM/DI/0282018
Record Dates: First submitted 2023-09-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Vitamin D Deficiency; 25-Hydroxyvitamin D3 Deficiency, Selective
Keywords: Vitamin D3; enhanced egg; Vitamin D3-enhanced egg; 25-Hydroxyvitamin D3 Deficiency; supplementation; Mexico; Children
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin D Hydroxylation-Deficient Rickets, Type 1B

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind field trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Two types of eggs. Control egg and fortified egg (vitamin D3-enhanced egg), only the researcher in charge of eggs production was not blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D3-enhanced egg (Experimental): The experimental group consumed an vitamin D3-enhanced egg (~ 400 IU). The randomization unit was the take care SEDESOL centers. All children in 3 day-care centers were given one vitamin D3-enhanced egg at breakfast, 3 times a week for 12 weeks (Monday, Wednesday and Friday).
  Interventions: Dietary Supplement: vitamin D-enhanced egg
- Control (Placebo Comparator): The control group consumed unfortified egg (~ 43 IU Vitamin D). The randomization unit was the 6 day-care centers (SEDESOL). All children in 3 day-care centers were given unfortified egg at breakfast, 3 times a week for 12 weeks (Monday, Wednesday and Friday).
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: vitamin D-enhanced egg — In our study, the vitamin D3-enhanced eggs were produced by hens that received 23,500 IU of vitamin D3 per kg of feed. Which does not confer them any harm or danger of intoxication. This experiment was carried out at the Center for Teaching, Research and Extension in Poultry Production (CEIEPAv, FMVZ-UNAM) and lasted 40 weeks.
  This ensured that the hens eggs were enhanced with vitamin D achieving a final concentration of approximately 400 IU of vitamin D
  Arms: vitamin D3-enhanced egg
Other: Control — Unfortified eggs were used for the control group with a concentration of approximately 43 IU of vitamin D
  Arms: Control

SUMMARY:
This is double-blind, controlled fiel trial, to compare fortified egg with D3-or 25(OH)D3 and non-fortified eggs in healthy preschool-age children 12 to 60 months of age, affiliated to day-care centers at Secretaria de Desarrollo Social (SEDESOL).

The study aims to answer are:

1. to evaluate the efficacy of fortified egg with vitamian D3 on serum concentrations of 25-hydroxyvitamin D3
2. and to evaluate parathyroid hormone (PTH) in children aged 12 to 60 months of age.

   * Children would be given for breakfast fortified egg/non-foritfied egg three times per week for 12 weeks.
   * Blood samples will be taken at baseline and at the end of study.
   * Anthropometric meassurements weight /height will be taken at baseline and at end of study.

DETAILED DESCRIPTION:
1. Vitamin D functions:

   Vitamin D (VD) is a fat-soluble vitamin. Its main function is to maintain optimal levels of calcium and phosphorus in the body; it also helps in neuromuscular transmission and bone mineralization, important in bone health and growth in children. There are VD receptors in bone, bone marrow, adipose tissue, adrenal, brain, stomach, small intestine, colon, pancreas, liver, lung, muscle, activated B and T lymphocytes, and in other organs, tissues, and cells. For this reason, various functions are assumed. VD serum concentrations above 75 mmol/l (30 ng/ml) have been shown to keep cell growth under control and prevent cells from becoming autonomous and malignant.
2. Prevalences of vitamin D deficiencies and insufficiency:

   Worldwide, a high proportion of children, youth, and middle-aged adults are deficient in Vitamin D. It has been estimated that about one billion people in the world may be deficient in Vitamin D.

   In Latin America, only Mexico has representative population data on vitamin D deficiency. Recently it has been documented that the deficiency and insufficiency of Vitamin D are a public health problem in Mexico. In a national representative sample of 6,827 children aged 1 to 11 years who participated in the 2012 National Health and Nutrition Survey (ENSANUT), the prevalence of Vitamin D deficiency was 33% (25-OH-D <50 nmol/L), which means that there are 3 million children with Vitamin D deficiency in Mexico. On the other hand, insufficiency (25-OH-D of 50 <75 nmol/L) affects 56% of children. Likewise, it was found that less than 3% of children consume a supplement with Vitamin D.
3. Vitamin D intake recommendations in children:

   The current vitamin D intake recommendations made by the APP since 2008 (Wagner CL, 2008) for children aged 1 to 8 years is an Adequate Intake of 400-600 IU (10-15µg), and for the Tolerable Upper Intake Level it is suggested do not exceed 2500 IU (63µg) in the case of children from 1 to 3 years and 3000 IU (75µg) in children from 4 to 8 years.
4. Description of the study:

   A double-blind controlled cluster randomized field trial was developed.

   The participants were children from 6 day-care centers (SEDESOL) at Cuernavaca, Morelos, Mexico. The study sample had 275 children that completed the study (the protocol considered having at least 125 children in each treatment group), from 12 to 59 months, who attended 6 take care centers (SEDESOL), in Cuernavaca, Morelos.
5. Objective

   To evaluate the efficacy of the consumption of fortified eggs with Vitamin D3 on the serum concentrations of 25-OH-D in children aged 12 to 59 months who attend take care centers (SEDESOL)in Cuernavaca.
6. Treatment and control groups:

   The random assignments of the intervention group (fortified egg) and control group (unfortified egg) were done considering each day-care center as a unit of allocation.

   Three day-care centers were randomized to the intervention group and three to the control group. The study lasted 12 weeks.

   The treatment group consumed a fortified egg to provide 10 mcg of Vitamin D3 equivalent to 400 IU of Cholecalciferol, 3 times a week.

   The control group received unfortified egg (~ 43 IU Vitamin D) with the same frequency as the intervention group.
7. Main Outcomes:

   The main outcome outcome variables were the serum levels of 25-hydroxyvitamin D3 (25-OH-D3) The second main outcome was to evaluate the parathyroid hormone (PTH).

   Other Variables:

   Blood parameters were taken: total cholesterol, HDL cholesterol, triglycerides, glucose, and hemoglobin.

   Anthropometric measurements of weight, height, age.

   Morbidity (diarrhea, constipation and respiratory tract infections) was evaluated three times per week and recorded.

   Standardized personnel weight the egg consumed before and after breakfast with a food weighing scale.

   Mothers were asked about children's usual diet by two diet questionnaires : a 24-hour dietary recall and a food frequency questionnaire at baseline and at the end of the study.
8. Ethical considerations:

The protocol was submitted to he Research and Ethics Committee of the Medicine Research Division of the National Autonomous University of Mexico.The study was approved on May 8, 2018 with folio FM/DI/028/2018.

The children's mothers or guardians signed an informed consent letter.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex, from 12 to 59 months of age who attend take care SEDESOL centers
* Children who consume eggs within their usual diet at least 5 times per month
* Childrens whose parents or legal guardian agree to participate in the study and sign an informed consent letter

Exclusion Criteria:

* Children with an egg allergy
* Chldren with hypersensitivity to vitamin D
* Children who have taken vitamin D supplements in the past month

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Serum 25-OH-D | At baseline and at 12 weeks of intervention
  nmol/L

SECONDARY OUTCOMES:
Serum PTH | At baseline and at 12 weeks of intervention
  pcg/mL

OTHER OUTCOMES:
Insulin | At baseline and at 12 weeks of intervention
  ug/dL
Weight | At baseline and at 12 weeks of intervention
  kg
Height | At baseline and at 12 weeks of intervention
  cm
Total Cholesterol | At baseline and at 12 weeks of intervention
  mg/dL
Triglicerids | At baseline and at 12 weeks of intervention
  mg/dL
HDLc | At baseline and at 12 weeks of intervention
  mg/dL
Glucose | At baseline and at 12 weeks of intervention
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Mario E Flores Aldana, PhD, Principal Investigator — National Institute of Public Health, Mexico
Locations (1):
- Instituto Nacional de Salud Pública, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No